CLINICAL TRIAL: NCT07403435
Title: Short-course Radiotherapy Combined With Serplulimab and Chemotherapy as Neoadjuvant Treatment for Resectable Esophageal Squamous Cell Carcinoma: a Single-center, Open-label Phase II Clinical Trial
Brief Title: Short-course Radiotherapy Combined With Serplulimab and Chemotherapy as Neoadjuvant Treatment for Resectable ESCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT163
Record Dates: First submitted 2025-09-08; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Short-course radiotherapy; neoadjuvant; esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Albumin-Bound Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): PTV:1.5Gy Bid,5 days Serplulimab (300mg) + Albumin-bound paclitaxel + Cisplatin/Carboplatin, Q3W, 3cycles
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — Serplulimab (300mg) + Albumin-bound paclitaxel + Cisplatin/Carboplatin, Q3W, 3cycles
  Other Names: Albumin-bound paclitaxel; Cisplatin; Carboplatin

SUMMARY:
This study includes patients with resectable esophageal squamous cell carcinoma who will undergo local radiotherapy (PTV: 1.5Gy Bid, for 5 days), followed by neoadjuvant treatment with Serplulimab combined with cisplatin and paclitaxel for three cycles. Afterward, they will undergo surgery. Postoperatively, researchers will select adjuvant treatment plans based on the patients' conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed squamous cell carcinoma of the esophagus (ESCC) staged as cT1-2N+M0 and cT3NanyM0 (AJCC 8th edition);
2. Aged between 18-75 years;
3. ECOG performance status score of 0-1;
4. The following laboratory tests confirm that the bone marrow, liver and kidney functions meet the requirements for study participation

   1. Hemoglobin ≥90g/L; ANC≥1.5×10^9/L;platelet count ≥100×10^9/L (patients must not have received blood transfusion or growth factor support within 14 days of blood sample collection);
   2. ALT, AST ≤2.5*ULN; ALP ≤2.5*ULN;
   3. Serum total bilirubin <1.5*ULN
   4. Serum creatinine <1.5*ULN or estimated glomerular filtration rate (eGFR) ≥60ml/min/1.73m^2;
   5. Serum albumin ≥30g/L;
   6. INR or PT ≤1.5 *ULN, unless the patient is on anticoagulant therapy and the PT is within the expected therapeutic range; g. Activated partial thromboplastin time (APTT) ≤1.5 times ULN.
5. No severe concomitant diseases with a life expectancy of less than 5 years;
6. Voluntary and able to comply with the study protocol during the study period;
7. Provide written informed consent prior to entering the study, and the patient has been informed that they can withdraw from the study at any time without any loss.

Exclusion Criteria:

1. History of other malignancies in the past or concurrently, except for cured basal cell carcinoma of the skin and in situ cervical carcinoma; patients with small gastric stromal tumors and other tumors judged by the investigator to not affect the patient's life in the short term may be excluded;
2. Participation in other drug clinical trials within four weeks;
3. Patients with any active autoimmune disease or history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaryitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; asthma that was completely resolved in childhood and does not require any intervention in adulthood may be included; asthma requiring medical intervention with bronchodilators cannot be included);
4. Patients currently using immunosuppressants, or systemic corticosteroid therapy for immunosuppressive purposes (dose >10mg/day prednisone or other equivalent corticosteroids), and continued use within two weeks prior to enrollment;
5. Any active malignant tumor within two years, except for the specific cancer being studied in this trial and cured locally recurrent cancer (e.g., resected basal cell or squamous cell skin cancer, superficial bladder cancer, in situ cervical or breast carcinoma);
6. Patients with known central nervous system (CNS) metastasis or history of CNS metastasis at screening. For patients clinically suspected of CNS metastasis, a CT or MRI examination must be performed within 28 days before treatment to rule out CNS metastasis;
7. History of unstable angina; newly diagnosed angina within three months before screening or myocardial infarction event within six months before screening; arrhythmia (including QTcF: males ≥450 ms, females ≥470 ms) requiring long-term antiarrhythmic medication and New York Heart Association class ≥II heart failure;
8. Urine routine indicating proteinuria ≥++ and confirmed 24-hour urinary protein >1.0 g;
9. For female subjects: should be surgically sterilized, postmenopausal patients, or agree to use a medically recognized contraceptive method during the study treatment period and for six months after the end of the study treatment; serum or urine pregnancy test must be negative within seven days before study enrollment, and must not be lactating. For male subjects: should be surgically sterilized, or agree to use a medically recognized contraceptive method during the study treatment period and for six months after the end of the study treatment;
10. Patients who have undergone liver transplantation;
11. Infectious pneumonia, non-infectious pneumonia, interstitial pneumonia, and other patients requiring the use of corticosteroids;
12. History of chronic autoimmune diseases, such as systemic lupus erythematosus;
13. History of inflammatory bowel diseases such as ulcerative colitis, Crohn's disease, and history of chronic diarrheal diseases such as irritable bowel syndrome;
14. History of sarcoidosis or tuberculosis;
15. Active hepatitis B, hepatitis C, and HIV infection;
16. Untreated active syphilis;
17. History of substance abuse with psychotropic drugs and unable to quit or with psychiatric disorders;
18. Pleural effusion or ascites with clinical symptoms requiring clinical intervention;
19. History of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
20. According to the investigator's judgment, there are serious concomitant diseases that endanger patient safety or affect the patient's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
pCR（Pathological Complete Response） | within 14 working days after operation
  Definition of pathology complete response is "no cancer cell, including lympho nodes"

SECONDARY OUTCOMES:
MPR（Major Pathological Remission rate） | within 14 working days after operation
  The residual tumor after neoadjuvant treatment ≤ 10% residual tumor lesion in surgical specimen compared to baseline.
ORR（Objective Response Rate） | 3-4 weeks after the last cycle of neoadjuvant treatment
  The Objective Response Rate (ORR) will be defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) (RECIST V1.1)
Rate of R0 resection | within 14 working days after operation
  Measure the rate of R0 resection with all margins microscopically clear.
EFS (Events Free Survival) | The date from the beginning of randomization to the date of first record. 5 years EFS
  The time from the start of treatment until any of the following events occur: any disease progression that prevents surgery, postoperative disease progression or recurrence, or death due to any cause
Safety assessment | From the first dose of study drug up to 30 days after last dose of any component of treatment or surgery or the initiation of subsequent anticancer therapy, whichever occurred first. Up to approximately 9 months.
  Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No